CLINICAL TRIAL: NCT03157908
Title: A Pilot Study to Assess the Acceptability and Feasibility of a Smartphone App to Improve Retention in Postpartum HIV Care in South Africa
Brief Title: CareConekta: A Pilot Study of a Smartphone App in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Kate Clouse, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 170510
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: HIV/AIDS
Keywords: South Africa; Retention in care; Pregnancy; Mobile health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone app (Experimental): All participants in this pilot study will install the smartphone app for testing
  Interventions: Device: CareConekta

INTERVENTIONS:
Device: CareConekta — CareConekta is a smartphone app developed in parallel with a series of focus group discussions that uses global positioning system (GPS) data to identify the user's location to meet two primary functions: (1) to allow the participant to locate ART facilities in South Africa that are near her current location, and (2) to trace mobility prospectively.

SUMMARY:
Population mobility is frequent in South Africa and disrupts the continuity of HIV care. Postpartum, HIV-positive women are at elevated risk of dropping out of HIV care and are highly mobile. This pilot study aims to engage peripartum, HIV-positive women as potential users to evaluate a novel smartphone application to assist these women with linkage to new HIV facilities and prospectively describe the mobility of this population.

DETAILED DESCRIPTION:
South Africa is home to the world's largest antiretroviral therapy (ART) program, but sustaining high retention along the HIV care continuum has proven challenging in the country and throughout the wider region. Population mobility is frequent in South Africa and mobility likely disrupts retention in HIV care. In the absence of a facility-linked national electronic health data system, clinic switching as unreported transfers also obscures the true magnitude of loss to follow-up, hindering national evaluation efforts. Postpartum women in South Africa are known to be at high risk of dropping out of HIV care after delivery and are frequently mobile, partly due to cultural traditions of returning to one's rural home after giving birth. To address these challenges to retention in care, the investigators will enroll 30 peripartum, HIV-positive women as potential users to assess the acceptability and feasibility of deploying in a real-world setting a novel mHealth application to improve retention in HIV care. The app will operate on users' own smartphones and will serve two primary functions: 1) as a service tool to inform postpartum, HIV-positive women of ART services in their area so that they may access continued HIV care, even while traveling, and 2) as a research tool to prospectively characterize travel and mobility patterns of these women. During this pilot study, women will be passively followed for 90 days following app installation at enrollment. After 90 days, they will be interviewed to determine acceptability and feasibility, and electronic user data will be analyzed. This information will be used to develop an app poised for nationwide adoption. The research team comprises leaders in the study of HIV implementation science, maternal/child health and biomedical informatics, with experience designing effective mobile health (mHealth) interventions in low-resources settings. This pilot study aims to engage potential users to test a smartphone application that both improves linkage to HIV care and provides essential research data to inform future health system strengthening efforts.

ELIGIBILITY:
Inclusion Criteria:

* Willing to enroll and provide written informed consent
* ≥18 years old
* HIV-positive
* Pregnant (>36 weeks gestation)
* Able to read basic written English
* Currently own a smartphone that meets the technical requirements
* Willing to opt-in to installation of the app on her personal phone and to mobility tracking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Feasibility questionnaire | 3 months
  Feasibility will be assessed via a face-to-face questionnaire to address the following questions:
  * What proportion of women eligible to participate chooses to participate in the study?
  * Are participants able to install the app on their phones?
  * How does real-world access to the internet affect the use of the app?
  * When is the optimal time for the participant to receive a notification?
  * How many notifications are sent?
  * What unexpected problems occurred?
  * What are the general usage patterns of the app?
Acceptability questionnaire | 3 months
  Acceptability will be assessed via a face-to-face questionnaire to address the following questions:
  * Do women find the app helpful?
  * How frequently do women engage with the app and under what circumstances?
  * Do women report that they think such an app should be offered to other pregnant women? What about to non-pregnant adults?
  * Are there other services that participants would like to see included on future version of the app?
  * Do women like the notifications?

SECONDARY OUTCOMES:
Medical record review to assess potential efficacy | 3 months
  The investigators will assess paper and electronic medical records to assess if the receipt of a notification results in linkage to a facility, as recorded through self-report and patient records.
Spatial analysis of GPS data | 3 months
  The investigators will analyze the GPS data collected in during the pilot study to determine the characteristics of peripartum women's mobility patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Clouse, PhD, MPH, Principal Investigator — Vanderbilt University Medical Center; Tamsin K Phillips, MPH, Principal Investigator — University of Cape Town
Locations (1):
- Gugulethu Community Health Centre, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No